CLINICAL TRIAL: NCT05263713
Title: Aesthetic Outcome of Running Subcuticular Suture Versus Running Horizontal Mattress Suture Closure of Linear Wounds on the Trunk and Extremities: a Randomized Evaluator Blinded Split Wound Comparative Effectiveness Trial
Brief Title: Aesthetic Outcome of Running Subcuticular Suture Versus Running Horizontal Mattress Suture Closure of Linear Wounds on the Trunk and Extremities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: 1813469
Record Dates: First submitted 2021-11-30; First posted 2022-03-03 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Wound of Skin; Scar
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Intervention Model Description: At the follow-up visit, two blinded observers will record their scores independently using the POSAS instrument.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Running Horizontal Mattress (Experimental): Half of the wound is repaired with running horizontal mattress sutures
  Interventions: Other: Suture Closure of Linear Wounds
- Running Subcuticular Suture (Experimental): Half of the wound is repaired with running subcuticular sutures
  Interventions: Other: Suture Closure of Linear Wounds

INTERVENTIONS:
Other: Suture Closure of Linear Wounds — Half of the wound is repaired with running subcuticular sutures and the other half is repaired with running horizontal mattress sutures.

SUMMARY:
The purpose of this study is to determine whether the use of running subcuticular suture versus running horizontal mattress suture for the repair of cutaneous linear wounds on the trunk and extremities affects aesthetic outcomes. The study team will use a split wound model, where half of the wound is repaired with running subcuticular sutures and the other half is repaired with running horizontal mattress sutures. Three-months post-surgery, the scar will be evaluated via the patient observer scar assessment scale (POSAS), a validated scar instrument, as well as the trace-to-tape method, an objective outcome measure for linear postoperative scars. Any adverse events will also be recorded.

DETAILED DESCRIPTION:
Sutures are the standard of care in repairing cutaneous wounds. The majority of surgical reconstructions following a Mohs micrographic surgery and standard surgical excisions require two layers of sutures: a deep (subcutaneous) layer and a superficial (cuticular) layer. Given the overall lack of evidence in the literature, the choice of suturing technique is largely dependent on the surgeon's preference.

This study aims to investigate whether the use of running subcuticular sutures, when compared to running horizontal mattress sutures, affects wound cosmesis on the trunk and extremities.

Both running subcuticular and horizontal mattress suture techniques have been favored by surgeons for differing reasons. With running subcuticular suture, epidermal puncture points are minimized. Thus, suture may be left in place for longer periods of time leading to improved wound healing and less risk of suture-track scars. A previous study by Alam et al found that running subcuticular suture had improved appearance as compared to running cuticular suture. In contrast, the horizontal mattress suture is useful to redistribution wound tension and evert wound edges, which is felt to improve aesthetic surgical outcomes as well. Moody et al showed that when compared to running cuticular suture, a running horizontal mattress suture led to a smoother and flatter scar.

However, while there have been studies comparing and finding superiority of both the subcuticular running suture and running horizontal mattress suture compared to the running cuticular suture, these two techniques (namely, subcuticular running and running horizontal mattress) have not been directly compared to each other. We hope that our study will provide new insight into this aspect of cutaneous surgery.

This is a single center, randomized, evaluator blind, split wound study.

After screening and informed consent, demographic data will be collected including date of birth, race, gender and medical record number.

The patient's wound will be labeled A if it is on the left or superior side of the investigator and B if it is on the right or inferior side. A predetermined, concealed randomization number will be obtained from the redcap randomization module, which will specify how side A is to be treated. Side B will be treated the opposite way as A. Side A will always be closed first. Prior to placement of the cutaneous sutures, both sides of the wound will be sutured together with a subcutaneous (bottom) layer of stitches, as is the standard of care. A digital image of the wound before and after the epidermal closure will be obtained; these may be used in scientific talks and/or for publication purposes. Treatment assignment, wound length, demographic data, and digital images will be recorded within the redcap database. Follow-up assessment will be scheduled for three months following the procedure, with a one-month window before or after that time if the patient cannot return at precisely three months.

At the follow-up visit, two blinded observers will record their scores independently using the POSAS instrument. The mean scar width will also be determined using the trace-to-tape method. If one half of the scar has more associated erythema, that will be recorded. The patient part of the instrument will be independently recorded. Digital images will then be obtained again, which may be used for scientific meeting presentation and/or publication purposes.

ELIGIBILITY:
All patients scheduled for cutaneous surgical procedures with one of the study investigators at the UC Davis Dermatology Clinic will be screened for eligibility.

Inclusion Criteria:

* 18 years of age or older
* Able to give informed consent themselves
* Patient scheduled for cutaneous surgical procedure on the trunk or extremities with predicted primary closure
* Willing to return for follow up visit

Exclusion Criteria:

* Incarceration
* Under 18 years of age
* Pregnant Women
* Wounds with predicted closure length less than 3 cm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Scar Assessment as measured by Patient Observer Scar Assessment Score (POSAS) | 3 months
  The primary endpoint will be the score of two blinded reviewers independently using the POSAS assessment. The observer scale of the POSAS consists of six items (vascularity, pigmentation, thickness, relief, pliability, and surface area). All items are scored on a scale ranging from 1 ("like normal skin") to 10 ("worst scar imaginable"). The sum of the six items results in a total score of the POSAS observer scale. Furthermore, an overall opinion is scored on a scale ranging from 1 to 10. All parameters should preferably be compared to normal skin on a comparable anatomic location.
Width of Scar as measured using Trace-to-Tape Method | 3 months
  The trace-to-tape method is an objective measure for linear postoperative scars. The mean scar width will be determined using the trace-to-tape method. The surface area of the scar will be collected by tracing the scar with a water-based gel pen. While still wet, the gel residue will be lifted from the skin with clear packing tape and transferred on a sheet of paper.

SECONDARY OUTCOMES:
Complications or Adverse Events from Treatment | 3 months
  For example, if one half of the scar has more associated erythema, as measured using the Trace-to-Tape method, then it will be recorded. Other complications from the treatment will also be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Davis, Sacramento, California, United States

REFERENCES:
- [Background] Robinson, J. Surgery of the Skin. New York, NY: Elsevier. 2014.
- [Background] Alam M, Posten W, Martini MC, Wrone DA, Rademaker AW. Aesthetic and functional efficacy of subcuticular running epidermal closures of the trunk and extremity: a rater-blinded randomized control trial. Arch Dermatol. 2006 Oct;142(10):1272-8. doi: 10.1001/archderm.142.10.1272. PMID 17043181
- [Background] Moody BR, McCarthy JE, Linder J, Hruza GJ. Enhanced cosmetic outcome with running horizontal mattress sutures. Dermatol Surg. 2005 Oct;31(10):1313-6. doi: 10.1111/j.1524-4725.2005.31209. PMID 16188185